CLINICAL TRIAL: NCT07185646
Title: The Second Xiangya Hospital of Central South University
Brief Title: Mechanistic Study of SPARC-Mediated Regulation of Neutrophil Extracellular Trap Formation in the Brain Metastatic Microenvironment of Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yu Zhou, Assistant Researcher, Second Xiangya Hospital of Central South University
Other Study IDs: 32200747
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Neuro-Oncology; MRI Imaging; Tumor Immune Microenvironment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to investigate the characteristics of the tumor microenvironment in patients with brain tumors using multi-modal magnetic resonance imaging (MRI). The primary research question it aims to address is:

• Can multi-modal MRI effectively characterize features of the immune microenvironment in brain tumor patients?

Participants:

Eligible participants who have been diagnosed with a brain tumor will undergo multi-modal MRI scans for detailed assessment of tumor microenvironment features.

ELIGIBILITY:
Inclusion Criteria:

1. conventional MRI revealed intracranial space-occupying lesions and suspected high-grade gliomas, brain metastases and meningiomas；
2. It is planned to perform a brain tumor resection surgery in this institution.

Exclusion Criteria:

1. other CNS diseases in addition to brain tumors;
2. pathologically confirmed brain tumors not belonging to any of the three selected types;
3. contraindications to the use of gadolinium contrast, including hypersensitivity to contrast agents, renal dysfunction, pregnancy or lactation;
4. contraindications to MRI;
5. poor image quality unsuitable for subsequent analyses;
6. age younger than 18 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Progression-Free Survival | 6months，12months，24months
  Postoperative Progression-Free Survival is defined as the time interval from the date of surgical intervention until the first occurrence of either documented disease progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No